CLINICAL TRIAL: NCT07238790
Title: A Phase 1 Study to Evaluate the Safety of a Complex Gut Bacterial Consortium (MITI 001) for the Treatment of Irritable Bowel Syndrome With Diarrhea
Brief Title: Use of A Complex Gut Bacterial Consortium (MITI 001) for the Treatment of Irritable Bowel Syndrome With Diarrhea
Acronym: CURE-IBS-D
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Spencer, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 82277; 31936 (Registry Identifier: FDA IND application number)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: IBS (Irritable Bowel Syndrome); Diarrhea
Keywords: IBS with Diarrhea Predominance (IBS-D)
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention arm (MITI-001) (Experimental): Dosed with MITI-001
  Interventions: Drug: MITI-001 administration

INTERVENTIONS:
Drug: MITI-001 administration — A complex gut bacterial community (MITI-001) will be given endoscopically and orally

SUMMARY:
While the pathophysiology of diarrhea-predominant irritable bowel syndrome (IBS-D) is complex and heterogeneous, dysbiosis of the gut microbiome is frequently observed, suggesting that a substantial subset of patients with irritable bowel syndrome (IBS) have symptoms that are initiated and/or perpetuated by a microbiome dysfunction. Successful randomized controlled trials (RCT) for IBS-D (Ford 2018; Black 2022) leveraging microbiome-targeted therapies (antibiotics or low microbiome fermentation diets) suggest the gut microbiome is at least partially involved in IBS symptoms. Furthermore, fecal microbiota transplantation (FMT) for patients with IBS-D has demonstrated promising results (El-Salhy 2020), supporting the possibility that altering the microbiome composition could ameliorate IBS-D symptoms.

MITI-001 is a transplantable gut bacterial community composed of 157 live bacterial strains, encompassing 79 genera of commensal bacteria, that have been isolated from healthy donor stool, purified, and banked. The hypothesis of the proposed research is that MITI-001 can target the pathophysiologic lesion in a subset of IBS-D patients, restore the altered microbial metabolic process, and thus alleviate IBS-D symptoms.

DETAILED DESCRIPTION:
MITI-001 has not yet been tested in humans. However, several RCTs support the role of the gut microbiome in IBS-D pathogenesis. These include trials involving non-absorbable antibiotics (e.g., rifaximin) and low-fermentation diets (Ford 2018; Black 2022), which have demonstrated symptom improvement. FMT has also shown promising efficacy in IBS-D (El-Salhy 2020), particularly when pre-treatment with antibiotics and/or bowel lavage was used to deplete the resident microbiota (Ianiro 2022; Zhang 2024). These findings highlight the need for introduction of a complete microbial ecosystem, rather than enrichment of isolated species, to achieve stable engraftment and functional restoration.

MITI-001 is uniquely designed to address both the compositional and functional deficiencies observed in a subset of IBS-D patients. It contains bacterial species capable of bile acid metabolism (bile salt hydrolase and 7α-dehydroxylation), potentially restoring the physiological bile acid pool. Given that isolated supplementation of missing species has been insufficient due to niche occupancy and dysbiosis, a complete defined community is required.

Prior clinical trials have demonstrated a consistent signal suggesting efficacy of FMT (Halkjær 2018; El-Salhy 2020; Aroniadis 2019; Lahtinen 2020; Johnsen 2018; Johnsen 2020; Holvoet 2021). Trials with high-dose endoscopic delivery have been the most successful and support the approach to be used in the proposed study (El-Salhy 2020; Holvoet 2021).

The planned Phase 1, open-label, single-arm, single-center study will evaluate MITI-001, a consortium of 157 live bacterial strains, as a possible treatment for participants with IBS-D. Each study participant will undergo screening assessments, a four-week observation period to quantify baseline symptoms, a nine-day treatment period, and a three-month follow-up period.

During the treatment period, participants will be pre-treated for five consecutive days with a combination of oral broad-spectrum antibiotics (vancomycin, metronidazole, and ciprofloxacin) to decrease the load of existing microbial colonists. One day prior to the first dose of MITI-001, oral antibiotic pre-medication will be stopped, and an orally administered bowel lavage will be performed. On Day 1, one dose of MITI-001 will be administered endoscopically to the duodenum (via esophagogastroduodenoscopy) and one dose will be administered to the ileum/distal colon (via colonoscopy). Participants will then self-administer MITI-001 orally twice daily on Days 2 to 4.

During the follow-up period, participants will have an in-person visit on Day 30 and virtual visits on Days 60 and 90 to monitor symptoms over time and collect stool samples for measurement of engraftment and bile acid composition. Throughout the study, participants will provide information about prior and concomitant medications and adverse events (AEs) via regular telephone or other virtual contacts with the site. A participant diary will be used to collect diet information and symptoms, as well as to administer questionnaires. Stool and urine samples will also be collected by the participant at home and delivered to the site.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years inclusive at the time of signing the informed consent.
2. Diagnosis of IBS-D according to the Rome IV criteria (Lacy 2017).
3. At least 1 of the following measures of microbiome dysfunction:

   1. Primary bile acid proportion ≥ 12% in stool samples, or
   2. Positive hydrogen breath test (with either glucose or lactulose substrate) (Rezaie 2017)
4. Normal C-reactive protein level
5. Gallbladder intact
6. Willing to use appropriate contraception during the treatment period and for one week after the last study visit.

   * Male participants with partners who are women of childbearing potential (WOCBP): Appropriate contraception includes condoms or other means considered adequate by the responsible Investigator.
   * Female participants who are WOCBP: Appropriate contraception includes condoms, an intrauterine device, hormonal contraception, or other means considered adequate by the responsible Investigator.
7. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol.
8. Able to tolerate the planned course of antibiotics, EGD, and colonoscopy with bowel lavage.

Exclusion Criteria:

1. Inflammatory bowel disease
2. Untreated enteric infections
3. History of gastrointestinal (GI) surgery: All participants with GI surgeries below the pylorus will be excluded from this study. This includes participants with a history of colectomy, segmental colonic resection, and small bowel resections.
4. Documented severe gastroparesis
5. Active intestinal obstruction
6. Dysphagia (oropharyngeal, esophageal, functional, or neuromuscular)
7. History of recurrent aspiration episodes
8. Any conditions associated with a high risk of bleeding, including but not limited to coagulopathy/bleeding disorder, severe liver disease, active or recent GI bleeding, or recent abdominal or other GI surgery
9. Active diagnosis of major depressive disorder
10. Severe immunodeficiency, inherited or acquired (e.g., human immunodeficiency virus, active chemotherapy or immunosuppressive medications [including steroids, biologic therapy, or bone marrow suppressive agent], or radiation therapy)
11. Any other significant medical condition that could confound or interfere with evaluation of safety or tolerability or prevent compliance with the study protocol at the discretion of the Investigator
12. Active antibiotic use (except protocol-specified antibiotics)
13. Active treatment with high levels of immunosuppressive therapies (active chemotherapy or immunosuppressive medications [including steroids, biologic therapies, or bone marrow suppressive agents], or radiation therapy)
14. Active anticoagulant or antiplatelet therapy, or use of other medications associated with a high risk of bleeding within 48 hours prior to endoscopy on Day 1
15. Use of a probiotic within one month prior to dosing of MITI-001 on Day 1
16. Simultaneous participation in another interventional clinical trial
17. Renal insufficiency (estimated glomerular filtration rate < 50 mL/min)
18. Absolute neutrophil count < 1000 μL, platelet count < 50 × 109/L, or hemoglobin level < 6.5 g/dL
19. Pregnant, breastfeeding, or planning pregnancy during the study period
20. Active drug or alcohol use disorder
21. Known allergy or anaphylaxis to vancomycin, metronidazole, ciprofloxacin, or polyethylene glycol
22. Inability to comply with research requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Determine the safety of MITI-001 in the participant population | up to 90 days
  Incidence of MITI-001-related adverse events

SECONDARY OUTCOMES:
Assess the ability of MITI-001 to restore microbial metabolic function: secondary bile acid metabolism and hydrogen consumption | Day 30 and Day 90
  * Restoration of metabolic normality (i.e., production of DCA and LCA, consumption of hydrogen)
  * Engraftment of bai (bile acid-inducible) operon-positive organism(s) measured via metagenomic analysis
  * Primary bile acid proportion < 12% in stool
Adequate relief of IBS-D symptoms | Day 30
  • Composite endpoint consisting of:
  * 50% or greater reduction in the number of days per week with stools of BSS types 6 or 7
  * 30% reduction in the weekly average of the worst daily abdominal pain, for at least 50% of the treatment weeks

OTHER OUTCOMES:
Determine whether restoration of microbial metabolic function leads to a reduction in IBS symptom burden in participants | up to 90 days
  IBS symptom burden as measured by:
  * IBS-SSS
  * Rome IV Questionnaire
  * BSS
  * Abdominal Bloating and Distension Pictogram
  * Gastrointestinal Symptom Rating Scale
  * IBS-QOL Survey
Measure the extent of engraftment at the taxonomic and cellular level | one week after last dose of MITI-001
  Percent of participants showing engraftment of > 30 strains from MITI-001 measured one week after the last dose of MITI-001
Measure the durability of engraftment and community stability over time | 90 days
  Percent of participants showing engraftment of > 15 strains from MITI-001 measured 90 days after the last dose of MITI-001

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fischbach, PhD, Study Director — Stanford University; Sean P Spencer, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Digestive Health Clinic, Redwood City, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No